CLINICAL TRIAL: NCT03619551
Title: A Randomized Trial of Low Versus Moderate Exposure Busulfan for Infants With Severe Combined Immunodeficiency (SCID) Receiving TCRαβ+/CD19+ Depleted Transplantation: A Phase II Study by the Primary Immune Deficiency Treatment Consortium (PIDTC) and Pediatric Blood and Marrow Transplant Consortium (PBMTC)
Brief Title: Conditioning SCID Infants Diagnosed Early
Acronym: CSIDE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBMTC NMD1801
Record Dates: First submitted 2018-07-16; First posted 2018-08-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: SCID
MeSH Terms: interventions — Busulfan

STUDY DESIGN:
Intervention Model Description: Randomization will be performed after eligibility is confirmed. Randomization between the two busulfan dose levels will be done separately in each genotype stratum, using permuted blocks. Randomization will be stratified further by donor type (Haploidentical related vs. Matched Unrelated Donor).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Low Dose Busulfan (Experimental): Busulfan based preparative regimen targeted at area-under-the-curve (cAUC) exposure of 25-35 mg*h/L .
  Randomization between the two dose levels will be done separately in each genotype stratum (RAG1/RAG2 and IL2RG/JAK3), using permuted blocks.
  Interventions: Drug: Busulfan; Device: Cell processing for TCRαβ+/CD19+ depletion
- Medium Dose Busulfan (Experimental): Busulfan based preparative regimen targeted at area-under-the-curve (cAUC) exposure of 55-65 mg*h/L.
  Randomization between the two dose levels will be done separately in each genotype stratum (RAG1/RAG2 and IL2RG/JAK3), using permuted blocks.
  Interventions: Drug: Busulfan; Device: Cell processing for TCRαβ+/CD19+ depletion

INTERVENTIONS:
Drug: Busulfan — Randomization between low and medium doses of busulfan for TCR αβ+/CD19+ depleted haploidentical related and unrelated donor HCT.
Device: Cell processing for TCRαβ+/CD19+ depletion — T-cells and B-cells will be removed from the stem cells collected from the donor by an investigational process called alpha-beta CD3+/CD19+ t-cell depletion using a device called CliniMACS® prior to recipient infusion, hopefully minimizing the risk of significant graft vs. host disease (GVHD) or lymphoproliferative disorder.
  Other Names: CliniMACS

SUMMARY:
The investigators want to study if lower doses of chemotherapy will help babies with SCID to achieve good immunity with less short and long-term risks of complications after transplantation. This trial identifies babies with types of immune deficiencies that are most likely to succeed with this approach and offers them transplant early in life before they get severe infections or later if their infections are under control. It includes only patients receiving unrelated or mismatched related donor transplants.

The study will test if patients receiving transplant using either a low dose busulfan or a medium dose busulfan will have immune recovery of both T and B cells, measured by the ability to respond to immunizations after transplant. The exact regimen depends on the subtype of SCID the patient has. Donors used for transplant must be unrelated or half-matched related (haploidentical) donors, and peripheral blood stem cells must be used. To minimize the chance of graft-versus-host disease (GVHD), the stem cells will have most, but not all, of the T cells removed, using a newer, experimental approach of a well-established technology. Once the stem cell transplant is completed, patients will be followed for 3 years. Approximately 9-18 months after the transplant, vaccinations will be administered, and a blood test measuring whether your child's body has responded to the vaccine will be collected.

DETAILED DESCRIPTION:
This is a prospective, multicenter, phase II, open-label study of two reduced busulfan dose levels in newborns identified at birth with SCID of appropriate genotype/phenotype and clinical status, undergoing either haploidentical related or well-matched unrelated donor TCRαβ+/CD19+ depleted HCT. Subjects will be enrolled on either of 2 strata according to genotype (defects of cytokine receptor function i.e. IL2RG or JAK3 and defects of receptor recombination i.e. RAG1 or RAG2). Thus up to 32 subjects on each of 2 strata or 64 subjects total would be enrolled over 4 years with 3 years follow-up.

Patients with IL2RG/JAK3 would be randomized to receive busulfan targeted either to cumulative exposure of 25-35 mg*h/L or 55-65 mg*h/L with Thymoglobulin. Patients with RAG1/2 would be randomized to receive busulfan targeted to cumulative exposure of 25-35 mg*h/L or 55-65 mg*h/L, in conjunction with fludarabine, thiotepa and Thymoglobulin. Safety/feasibility of the novel TCR αβ+/CD19+ depleted allogeneic HCT strategy will be monitored on an ongoing basis using stopping rules for lack of neutrophil engraftment and other important short-term toxicities.

Donor selection would be determined clinically at the discretion of the treating clinicians at each site. Pharmacokinetic monitoring of busulfan exposure will be performed per local practices at CLIA-certified laboratories. Patients will receive busulfan and pharmacokinetic measurement to individualize dosing. Time-concentration data of the initial dose and subsequent doses will be reviewed centrally (Dr. Janel Long-Boyle) using a cloud-based application (InsightRx) to guide dose adjustment in real-time (Long-Boyle, Chan, Keizer, 2017, ASBMT Tandem abstract accepted). Clinical and laboratory data will be collected at defined time points over 3 years and entered in an electronic data capture system using study-specific case report forms. These data will be used to measure the outcomes including the primary outcome (cAUC of busulfan that promotes humoral immune reconstitution at 2 years post HCT with acceptable regimen-related toxicity at 42 days post HCT) and secondary outcomes (the quality of donor cell engraftment and immune function achieved in B and T cell compartments and survival). Mechanistic studies supporting the exploratory endpoints will be conducted centrally in designated laboratories.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with SCID, either typical or leaky or Omenn syndrome.

1. Typical SCID is defined as either of the following

   * Absence or very low number of T cells (CD3+ T cells <300/microliter AND no or very low T cell function (<10% of lower limit of normal) as measured by response to phytohemagglutinin OR
   * Presence of maternally derived T cells
2. Leaky SCID is defined as the following

   • Absence of maternally derived T cells

   • AND either one or both of the following (i, ii): i) <50% of lower limit of normal T cell function as measured by response to PHA OR <30% of lower limit of normal T cell function as measured by response to CD3 ii) Absent or <10% of lower limit of normal proliferative responses to candida and tetanus toxoid antigens (must document post vaccination or exposure for this criterion to apply)

   • AND at least two of the following (i through iii): i) CD3 T cells < 1500/microliter ii) >80% of CD3+ or CD4+ T cells are CD45RO+ AND/OR >80% of CD3+ or CD4+ T cells are CD62L negative AND/OR >50% of CD3+ or CD4+ T cells express HLA-DR (at < 4 years of age) AND/OR are oligoclonal T iii) Low TRECs and/or the percentage of CD4+/45RA+/CD31+ or CD4+/45RA+/CD62L+ cells is below the lower level of normal.
3. Omenn syndrome • Generalized skin rash

   * Maternal lymphocytes tested for and not detected.
   * >80% of CD3+ or CD4+ T cells are CD45RO+ AND/OR >80% of CD3+ or CD4+ T cells are CD62L negative AND/OR >50% of CD3+ or CD4+ T cells express HLA-DR (<2 years of age)
   * Absent or low (up to 30% lower limit of normal (LLN)) T cell proliferation to antigens (Candida, tetanus) to which the patient has been exposed IF: Proliferation to antigen was not performed, but at least 4 of the following 8 supportive criteria, at least one of which must be among those marked with an asterisk (*) below are present, the patient is eligible as Omenn Syndrome.

     1. Hepatomegaly
     2. Splenomegaly
     3. Lymphadenopathy
     4. Elevated IgE
     5. Elevated absolute eosinophil count
     6. *Oligoclonal T cells measured by CDR3 length or flow cytometry (upload report)
     7. *Proliferation to PHA is reduced to < 50% of lower limit of normal (LLN) or SI < 30
     8. *Low TRECs and/or percentage of CD4+/RA+ CD31+ or CD4+/RA+ CD62L+ cells below the lower level of normal

     2. Documented mutation in one of the following SCID-related genes

a. Cytokine receptor defects (IL2RG, JAK3) b. T cell receptor rearrangement defects (RAG1, RAG2) 3. No available genotypically matched related donor (sibling) 4. Availability of a suitable donor and graft source

1. Haploidentical related mobilized peripheral blood cells
2. 9/10 or 10/10 allele matched (HLA-A, -B, -C, -DRB1, -DQB1) volunteer unrelated donor mobilized peripheral blood cells 5. Age 0 to 2 years at enrollment

Note: to ensure appropriate hepatic metabolism, age at time of busulfan start:

For IL2RG/JAK3: 8 weeks For RAG1/RAG2: 12 weeks

6. Adequate organ function defined as:

1. Cardiac:

   Left ventricular ejection fraction (LVEF) at rest ≥ 40% or, shortening fraction (SF) ≥ 26% by echocardiogram.
2. Hepatic:

   Total bilirubin < 3.0 x the upper limit of normal (ULN) for age (patients who have been diagnosed with Gilbert's Disease are allowed to exceed this limit) and AST and ALT < 5.0 x ULN for age.
3. Renal:

   GFR estimated by the updated Schwartz formula ≥ 90 mL/min/1.73 m2. If the estimated GFR is < 90 mL/min/1.73 m2, then renal function must be measured by 24-hour creatinine clearance or nuclear GFR, and must be > 50 mL/min/1.73 m2.
4. Pulmonary No need for supplemental oxygen and O2 saturation > 92% on room air at sea level (with lower levels allowed at higher elevations per established center standard of care).

Exclusion Criteria:

1. Presence of any serious life-threatening or opportunistic infection at time of enrollment and prior to the initiation of the preparative regimen. Serious infections as defined below that occur after enrollment must be reported immediately to the Study Coordinating Center, and enrollment will be put on hold until the infection resolves. Ideally enrolled subjects will not have had any infection. If patients have experienced infections, these must have resolved by the following definitions:

   a. Bacterial i. Positive culture from a sterile site (e.g. blood, CSF, etc.): Repeat culture(s) from same site must be negative and patient has completed appropriate course of antibacterial therapy (typically at least 10 days).

   ii. Tissue-based clinical infection (e.g. cellulitis): Complete resolution of clinical signs (e.g. erythema, tenderness, etc.) and patient has completed appropriate course of antibacterial therapy (typically at least 10 days).

   iii. Pneumonia, organism not identified by bronchoalveolar lavage: Complete resolution of clinical signs (e.g. tachypnea, oxygen requirement, etc.) and patient has completed appropriate course of antibacterial therapy (typically at least 10 days). If possible, radiographic resolution should also be demonstrated.

   b. Fungal i. Positive culture from a sterile site (e.g. blood, CSF, etc.): Repeat culture(s) from same site is negative and patient has completed appropriate course of antifungal therapy (typically at least 14 days). The patient may be continued on antifungal prophylaxis following completion of the treatment course.

   c. Pneumocystis i. Complete resolution of clinical signs (e.g. tachypnea, oxygen requirement, etc.) and patient has completed appropriate course of therapy (typically at least 21 days). If possible, radiographic resolution should also be demonstrated. The patient may be continued on prophylaxis following completion of the treatment course.

   d. Viral i. Viral PCRs from previously documented sites (blood, nasopharynx, CSF) must be re-tested and are negative.

   ii. If re-sampling a site is not clinically feasible (i.e. BAL fluid): Complete resolution of clinical signs (e.g. tachypnea, oxygen requirement, etc.). If possible, radiographic resolution should also be demonstrated.
2. Patients with HIV or HTLV I/II infection will be excluded.

Ages: 0 Years to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Vaccine specific antibody response | 2 years
  Humoral immune reconstitution by 2 years post HCT, defined by specific antibody response to tetanus toxoid. Criteria for evaluation of humoral immune response are the following:
  * Donor T cell chimerism ≥50%
  * B cell count ≥50 cells/microliter
  * IVIG independent for ≥12 weeks
  Subjects meeting the criteria receive 3 doses of tetanus toxoid at least 4 weeks apart, followed by measurement of tetanus titer at least 4-6 weeks after the 3rd dose. Those who achieve tetanus titer of ≥0.15 IU/ml after vaccination will meet the primary endpoint. Patients who have documented humoral immune response at a time prior to 2 years will be considered a success for the primary endpoint, while patients who do not have humoral immune response evaluated by 2 years will be considered failures for the primary endpoint.

SECONDARY OUTCOMES:
Immune Reconstitution | Up to 3 years
  * T cell immune reconstitution at 30 days, 60 days, 3 months, 6 months, 12 months, and 2 years post-HCT.
  * Naïve T cell generation and thymic output at 3 months, 6 months, 12 months and 2 years post-HCT.
  * Freedom from immunoglobulin substitution will be assessed on all patients at 9 months, 12 months, 2 years and 3 years post-HCT. Patients who have not received IVIG for at least 12 weeks at the time of assessment will be considered free from immunoglobulin substitution.
  * Tetanus responses on all patients who complete a trial of vaccination by additional timepoints of 12 months, 18 months and 3 years post-HCT.
  * Live vaccine responses on all patients who undergo trial of vaccination by 3 years post-HCT
Engraftment | Neutrophil Engraftment: 42 days post-HCT. Donor cell chimerism up to 2 years post-HCT.
  * Neutrophil engraftment will be assessed on all patients and defined as achieving an absolute neutrophil count of >500 cells/microliter for 3 consecutive days by day 42 post-HCT
  * Donor cell chimerism (whole blood, sorted CD3 (T-cell), CD19 (B-cell) and CD56 (NK cell) and granulocyte (CD15)) at 42 days, 3 months, 6 months, 12 months, and 2 years post-HCT. Absolute B cell, NK cell and granulocyte counts will be measured.
Overall Survival | 3 years
  Data to track overall survival will be collected at 1, 2 and 3 years post-HCT.
Event Free Survival | 3 years
  Data to track event free survival will be collected at 1, 2 and 3 years post-HCT. Events will be defined as 1) death from any cause, 2) rejection of the graft (T-cell and/or whole blood chimerism <5% donor), 3) graft failure necessitating a second HCT procedure from the same donor or a different donor, with or without conditioning, 4) DLI given for treatment of falling chimerism.
Acute graft-versus-host disease (aGVHD) | day 100 and 6 months post HCT
  Occurrence of acute (grade II-IV and grade III-IV) GVHD.
Chronic graft-versus-host disease (cGVHD) | 2 years post HCT
  Occurrence of chronic GVHD by 6 months, 12 months and 24 months post-HCT.
Post-HCT Complications | Up to 2 years post-HCT
  * Infections
  * Targeted regimen related toxicity (severe veno-occlusive disease of the liver, idiopathic pneumonitis syndrome)
  * Autoimmunity
Busulfan Pharmacokinetics | Pre-HCT
  Blood samples will be collected on busulfan dosing days 1 and 3 at 2.35, 4, 6 and 8 hours from the time of the start of the infusion. The results will be used to estimate individual exposure (AUC and cAUC).

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Yun Pai, MD, Study Chair — National Institutes of Health (NIH); Michael Pulsipher, MD, Study Chair — University of Utah
Locations (45):
- United States (42):
  - Univeristy of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona and Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCLA Center for Health Sciences, Los Angeles, California
  - Rady Children's Hospital, San Diego, San Diego, California
  - University of California San Francisco Medical Center - Peds, San Francisco, California
  - University of Colorado - Children's Hospital, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Shands HealthCare & University of Florida, Gainesville, Florida
  - University of Miami/Jackson Memorial Hospital, Miami, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Comer Children's Hospital/University of Chicago Medicine, Chicago, Illinois
  - Indiana University Hospital/Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Children's Hospital / LSUHSC, New Orleans, Louisiana
  - Dana Farber Cancer Institute - Peds, Boston, Massachusetts
  - The University of Michigan, Ann Arbor, Michigan
  - Helen DeVos Children's, Grand Rapids, Michigan
  - University of Minnesota Blood and Marrow Transplant Program - Pediatrics, Minneapolis, Minnesota
  - The Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Nebraska Medicine, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morgan Stanley Children's Hospital of New York-Presbyterian - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center - Peds, New York, New York
  - Cohen Children's Medical Center, Queens, New York
  - Westchester Medical Center, Valhalla, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center; Pediatric Blood and Marrow Transplant, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - Utah Blood and Marrow Transplant Program-Peds, Salt Lake City, Utah
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Montreal
  - The Hospital for Sick Children, Toronto, Ontario
  - Cancer Care Manitoba/University of Manitoba, Winnipeg, Winnipeg